CLINICAL TRIAL: NCT01045447
Title: A Trial Comparing Efficacy and Safety of NN5401 With Insulin Glargine, Both in Combination With Oral Antidiabetic Drugs in Subjects With Type 2 Diabetes (BOOST™ : INTENSIFY BASAL)
Brief Title: Comparison of NN5401 With Insulin Glargine, Both in Combination With Oral Antidiabetic Drugs, in Subjects With Type 2 Diabetes
Acronym: BOOST™
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN5401-3593; U1111-1111-7226 (Other: WHO); 2008-005767-34 (EudraCT Number)
Record Dates: First submitted 2010-01-08; First posted 2010-01-11 (Estimated); Results first posted 2015-11-18 (Estimated); Last update posted 2017-03-20 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin degludec, insulin aspart drug combination; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IDegAsp OD (Experimental)
  Interventions: Drug: insulin degludec/insulin aspart
- IGlar OD (Active Comparator)
  Interventions: Drug: insulin glargine

INTERVENTIONS:
Drug: insulin degludec/insulin aspart — Treat-to-target dose titration scheme, injected subcutaneously (under the skin) once daily with main meal. Dose was individually adjusted.
  Arms: IDegAsp OD
Drug: insulin glargine — Treat-to-target dose titration scheme, injected subcutaneously (under the skin) once daily. Dose was individually adjusted.
  Arms: IGlar OD

SUMMARY:
This trial is conducted in Africa, Asia, Europe and the United States of America (USA).

The aim of this clinical trial is to compare NN5401 (insulin degludec/insulin aspart) with insulin glargine in patients with type 2 diabetes inadequately controlled with insulin and oral anti-diabetic drugs (OADs). Subjects continued their ongoing treatment with OADs in the trial.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus (diagnosed clinically) for at least 6 months
* Treatment with basal insulin regimen (insulin detemir, insulin glargine or neutral protamine Hagedorn [NPH] insulin) once daily (OD), for at least 3 months
* Ongoing treatment with: metformin with or without other oral antidiabetic drugs (OADs) for at least 3 months prior to randomisation
* HbA1c 7.0-10.0 % (both inclusive) by central laboratory analysis
* BMI maximum 40.0 kg/m^2

Exclusion Criteria:

* Treatment with insulin regimens other than a basal insulin regimen (insulin detemir or insulin glargine or NPH insulin) OD within 3 months prior to Visit 1
* Treatment with glucagon-like peptide 1 (GLP-1) receptor agonists within 3 months prior to visit 1
* Current rosiglitazone users
* Cardiovascular disease, within the last 6 months prior to visit 1, defined as: stroke; decompensated heart failure New York Heart Association (NYHA) class III or IV; myocardial infarction; unstable angina pectoris; or coronary arterial bypass graft or angioplasty
* Uncontrolled treated/untreated severe hypertension (systolic blood pressure at least 180 millimetre (mm) mercury (Hg) and/or diastolic blood pressure at least 100 mmHg)
* Impaired liver function, defined as alanine aminotransferase (ALAT) at least 2.5 times upper limit of normal (one retest analysed at the central laboratory within a week of receipt of the result is permitted with the result of the last sample being conclusive)
* Pregnancy, breast-feeding, the intention of becoming pregnant or not using adequate contraceptive measures according to local requirements
* Cancer and medical history of cancer hereof (except basal cell skin cancer or squamous cell skin cancer)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 465 (Actual)
Dates: Start 2010-01; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (56):
- United States (22):
  - Novo Nordisk Investigational Site, Fresno, California
  - Novo Nordisk Investigational Site, Waterbury, Connecticut
  - Novo Nordisk Investigational Site, Boynton Beach, Florida
  - Novo Nordisk Investigational Site, Clearwater, Florida
  - Novo Nordisk Investigational Site, Jacksonville, Florida
  - Novo Nordisk Investigational Site, Kissimmee, Florida
  - Novo Nordisk Investigational Site, New Port Richey, Florida
  - Novo Nordisk Investigational Site, Orlando, Florida
  - Novo Nordisk Investigational Site, Pembroke Pines, Florida
  - Novo Nordisk Investigational Site, Tampa, Florida
  - Novo Nordisk Investigational Site, Atlanta, Georgia
  - Novo Nordisk Investigational Site, Des Moines, Iowa
  - Novo Nordisk Investigational Site, Baltimore, Maryland
  - Novo Nordisk Investigational Site, Hyattsville, Maryland
  - Novo Nordisk Investigational Site, Waltham, Massachusetts
  - Novo Nordisk Investigational Site, Southfield, Michigan
  - Novo Nordisk Investigational Site, Minneapolis, Minnesota
  - Novo Nordisk Investigational Site, Nashua, New Hampshire
  - Novo Nordisk Investigational Site, Albany, New York
  - Novo Nordisk Investigational Site, Statesville, North Carolina
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Round Rock, Texas
- Croatia (2):
  - Novo Nordisk Investigational Site, Osijek
  - Novo Nordisk Investigational Site, Rijeka
- France (7):
  - Novo Nordisk Investigational Site, Antibes
  - Novo Nordisk Investigational Site, Besançon
  - Novo Nordisk Investigational Site, Dax
  - Novo Nordisk Investigational Site, Paris
  - Novo Nordisk Investigational Site, Perpignan
  - Novo Nordisk Investigational Site, Saint-Herblain
  - Novo Nordisk Investigational Site, Sète
- India (8):
  - Novo Nordisk Investigational Site, Ahmedabad, Gujarat
  - Novo Nordisk Investigational Site, Bangalore, Karnataka
  - Novo Nordisk Investigational Site, Belagavi, Karnataka
  - Novo Nordisk Investigational Site, Mangalore, Karnataka
  - Novo Nordisk Investigational Site, Thiruvanathapuram, Kerala
  - Novo Nordisk Investigational Site, Pune, Maharashtra
  - Novo Nordisk Investigational Site, Bhubaneswar, Odisha
  - Novo Nordisk Investigational Site, Kanpur
- Poland (4):
  - Novo Nordisk Investigational Site, Gdansk
  - Novo Nordisk Investigational Site, Tychy
  - Novo Nordisk Investigational Site, Warsaw
  - Novo Nordisk Investigational Site, Wroclaw
- South Africa (2):
  - Novo Nordisk Investigational Site, Johannesburg, Gauteng
  - Novo Nordisk Investigational Site, Benoni
- South Korea (4):
  - Novo Nordisk Investigational Site, Busan
  - Novo Nordisk Investigational Site, Daegu
  - Novo Nordisk Investigational Site, Seoul
  - Novo Nordisk Investigational Site, Sungnam
- Sweden (5):
  - Novo Nordisk Investigational Site, Ängelholm
  - Novo Nordisk Investigational Site, Dalby
  - Novo Nordisk Investigational Site, Gothenburg
  - Novo Nordisk Investigational Site, Härnösand
  - Novo Nordisk Investigational Site, Stockholm
- Turkey (Türkiye) (2):
  - Novo Nordisk Investigational Site, Istanbul
  - Novo Nordisk Investigational Site, Kahramanmaraş

REFERENCES:
- [Result] Freemantle N, Mamdani M, Vilsboll T, Kongso JH, Kvist K, Bain SC. IDegLira Versus Alternative Intensification Strategies in Patients with Type 2 Diabetes Inadequately Controlled on Basal Insulin Therapy. Diabetes Ther. 2015 Dec;6(4):573-591. doi: 10.1007/s13300-015-0142-y. Epub 2015 Nov 18. PMID 26582052
- [Result] Kumar S, Jang HC, Demirag NG, Skjoth TV, Endahl L, Bode B. Efficacy and safety of once-daily insulin degludec/insulin aspart compared with once-daily insulin glargine in participants with Type 2 diabetes: a randomized, treat-to-target study. Diabet Med. 2017 Feb;34(2):180-188. doi: 10.1111/dme.13125. Epub 2016 Jul 28. PMID 27027878
- [Derived] Yang W, Akhtar S, Franek E, Haluzik M, Hirose T, Kalyanam B, Kar S, Wu T, Gogas Yavuz D, Unnikrishnan AG. Postprandial Glucose Excursions in Asian Versus Non-Asian Patients with Type 2 Diabetes: A Post Hoc Analysis of Baseline Data from Phase 3 Randomised Controlled Trials of IDegAsp. Diabetes Ther. 2022 Feb;13(2):311-323. doi: 10.1007/s13300-021-01196-7. Epub 2022 Jan 19. PMID 35044568
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 61 sites in 9 countries: Croatia (2 sites), France (4), India (8), Poland (4), South Africa (3), Republic of Korea (6), Sweden (5), Turkey (5) and United States of America (24).
Groups:
- IDegAsp OD: Insulin degludec/insulin aspart (IDegAsp) was given once daily (OD) subcutaneously (s.c.) with main evening meal or the largest meal of the day in combination with metformin±pioglitazone±DPP-4 inhibitor.
- IGlar OD: Insulin glargine (IGlar) was given once daily (OD) subcutaneously according to approved labelling in combination with metformin±pioglitazone±DPP-4. inhibitor.
Period: Overall Study
Arm/Group | IDegAsp OD | IGlar OD
Started | 232 | 233
Exposed | 230 (Two subjects withdrew prior to exposure to trial drug) | 233
Completed | 196 | 205
Not Completed | 36 | 28
Not completed — Adverse Event | 0 | 1
Not completed — Lack of Efficacy | 3 | 1
Not completed — Protocol Violation | 6 | 3
Not completed — Withdrawal Criteria | 10 | 10
Not completed — Unclassified | 17 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IDegAsp OD | IGlar OD | Total
Number analyzed (Participants) | 230 | 233 | 463
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.8 (9.5) | 58.4 (10.1) | 58.1 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95 | 106 | 201
  Male | 135 | 127 | 262
Glycosylated haemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin] | 8.3 (0.8) | 8.4 (1.0) | 8.3 (0.9)
Fasting plasma glucose (FPG) [Mean (Standard Deviation); unit: mmol/L] | 8.0 (2.5) | 7.8 (2.8) | 7.9 (2.7)

OUTCOME MEASURES:

1. Primary Outcome: Change in Glycosylated Haemoglobin (HbA1c)
Description: Change from baseline in HbA1c after 26 weeks of treatment.
Time Frame: Week 0, Week 26
Population: The full analysis set (FAS) included all randomised subjects and missing data was imputed using last observation carried forward (LOCF). Two subjects withdrew prior to exposure to trial drug, hence excluded from the FAS.
Measure: Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin
Arm/Group | IDegAsp OD | IGlar OD
Number analyzed (Participants) | 230 | 233
percentage of glycosylated haemoglobin | -0.98 (1.01) | -1.00 (1.06)

2. Secondary Outcome: Mean of 9-point Self Measured Plasma Glucose Profile (SMPG)
Description: Mean of SMPG after 26 weeks of treatment. Plasma glucose measured: before breakfast, 90 minutes after start of breakfast, before lunch, 90 minutes after start of lunch, before dinner, 90 minutes after start of dinner, bedtime, at 4 am and before breakfast.
Time Frame: Week 26
Population: The full analysis set (FAS) included all randomised subjects and missing data was imputed using last observation carried forward (LOCF). Two subjects withdrew prior to exposure to trial drug, hence excluded from the FAS. For 23 subjects all 9-point SMPG values were missing.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | IDegAsp OD | IGlar OD
Number analyzed (Participants) | 220 | 220
mmol/L | 8.1 (2.0) | 8.4 (2.0)

ADVERSE EVENTS:
Time Frame: The adverse events were collected in a time frame of 26 weeks + 7 days follow up.
Description: The safety analysis set included all subjects who received at least one dose of the investigational product or its comparator.
Arm/Group | IDegAsp OD | IGlar OD
Serious Adverse Events (participants affected / at risk) | 10/230 | 8/233
Other Adverse Events (participants affected / at risk) | 51/230 | 62/233
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDegAsp OD (N=230) | IGlar OD (N=233)
Angina pectoris (Cardiac disorders) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Haemorrhage (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDegAsp OD (N=230) | IGlar OD (N=233)
Diarrhoea (Gastrointestinal disorders) | 12 (15) | 13 (18)
Oedema peripheral (General disorders) | 5 (5) | 12 (12)
Nasopharyngitis (Infections and infestations) | 17 (21) | 18 (21)
Upper respiratory tract infection (Infections and infestations) | 11 (12) | 13 (13)
Headache (Nervous system disorders) | 20 (26) | 19 (26)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk maintains the right to be informed of any Investigator plans for publication and to review any scientific paper, presentation, communication or other information concerning the investigation described in this protocol. Any such communication must be submitted in writing to the Novo Nordisk trial manager prior to submission for comments. Comments will be given within four weeks from receipt of the planned communication.